CLINICAL TRIAL: NCT04099446
Title: A Non-Interventional Pilot Study to Explore the Skin Microbes in Skin Cancer Including Melanoma and Non-Melanoma
Brief Title: A Non-Interventional Pilot Study to Explore the Skin Microbes in Skin Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-003
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2021-04

CONDITIONS: Skin Cancer; Melanoma (Skin); Squamous Cell Carcinoma; Basal Cell Carcinoma; Microbiome
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Squamous Cell; Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Punch biopsies of skin from both cancerous and non-cancerous areas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Non-interventional — There is no intervention for this study

SUMMARY:
This study seeks to correlate microbial sequencing data from a punch biopsy in patients with skin cancer both melanoma and non-melanoma.

DETAILED DESCRIPTION:
The human Skin microbiome is a complex, interconnected web of microbes, living in a symbiotic relationship with their host. There are greater than ten times more bacteria on our bodies than there are human cells, all in a delicate and ever-changing balance to maintain a healthy skin microbiome. When this balance is disrupted, a condition known as dysbiosis, disease can occur. There is still a debate over whether dysbiosis is a cause of disease or a symptom of it. Naturally, since the microbiome has such a profound impact on human health, we want to study and learn as much about the microbiome as possible. By correlating this data with medical records for the patient's skin cancer, connections may begin to be drawn between organisms present in the microbiome of the skin microbiome, and skin cancer. Much like fingerprints, no microbiome is identical therefore the only chance we have at understanding disease is by looking at the skin microbiome and comparing the microorganisms on a patient with skin cancer biopsy and non-skin cancer biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years of age or older
* Diagnosis of skin cancer, both melanoma and non-melanoma
* Able/willing to have a skin punch biopsy in a non-cancerous location

Exclusion Criteria:

* Unable/unwilling to sign informed consent
* Inability to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 and older with a diagnosis of skin cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of Skin Microbiome to Cancer via Relative Abundance Found in Microbiome Sequencing | 1 year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the skin microbiome in both cancerous and non-cancerous areas. These data will then be compared to elucidate unique qualities of the microbiome in skin cancer.

SECONDARY OUTCOMES:
Validation of sequencing methods | 1 year
  To validate the sequencing methods used to generate microbiome data

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated, deidentified data will be made available to other researchers.